CLINICAL TRIAL: NCT01043263
Title: A Phase IIB, Randomized, Double-blind, Two-arm, Multi-center, Placebo-controlled, Study to Assess the Efficacy and Safety of EN3324 (Axomadol) in Subjects With Moderate to Severe Chronic Low Back Pain
Brief Title: Efficacy and Safety of EN3324 (Axomadol) in Subjects With Chronic Low Back Pain
Acronym: CLBP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EN3324-201
Record Dates: First submitted 2009-12-18; First posted 2010-01-06 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — axomadol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EN3324 (axomadol) (Experimental)
  Interventions: Drug: EN3324 (axomadol)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EN3324 (axomadol) — twice daily dosing
  Arms: EN3324 (axomadol)
Drug: Placebo — twice daily dosing
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of EN3324 (axomadol) in subjects with moderate to severe chronic low back pain

DETAILED DESCRIPTION:
A phase IIB, randomized, double-blind, two-arm, multi-center, placebo-controlled, study to assess the efficacy and safety of EN3324 (axomadol) in subjects with moderate to severe chronic low back pain

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Are females who are participating abstinence or using a medically acceptable form of contraception or have been post-menopausal, biologically sterile, or surgically sterile for more than 1 year.
* Have been on an unchanged regimen of analgesic medication for chronic low back pain on a daily basis for at least 3 months prior to screening; subjects taking opioids must not exceed total daily doses of 90mg oral morphine equivalent
* Have a history of moderate to severe CLBP

Exclusion Criteria:

* Have evidence of or a history of alcohol and/or drug abuse
* Have pain secondary to a confirmed or suspected neoplasm
* Intend to alter their physical therapy regimen during the study. Subjects who begin or end physical therapy (either home exercises or formal therapy sessions) 2 weeks prior to screening or during the study period will be excluded from the study
* Have a history or physical examination finding, which may confound pain-related data (e.g., fibromyalgia, radiculopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of EN3324 (axomadol) in subjects with moderate to severe CLBP. | Change from baseline [Day 0] to final visit [Day 112]

SECONDARY OUTCOMES:
To evaluate the safety, tolerability and efficacy of EN3324 (axomadol) in subjects with moderate to severe CLBP. | Change from baseline [Day 0] to final visit [Day 112]
To evaluate patient reported outcomes of EN3324 (axomadol) in subjects with moderate to severe CLBP. | Change from baseline [Day 0] to final visit [Day 112]

CONTACTS AND LOCATIONS:
Locations (59):
- United States (59):
  - Matthew Doust, MD, Phoenix, Arizona
  - Paradigm Clinical, Tucson, Arizona
  - Visions Clinical Research, Tucson, Arizona
  - Genova Clinical Research, Inc., Tucson, Arizona
  - Quality of Life Medical & Research Center, Tuscon, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Orange County Clinical Trials, Inc., Anaheim, California
  - Associated Pharmaceutical Research Center, Inc., Buena Park, California
  - Catalina Research Institute, LLC, Chino, California
  - Paradigm Clinical Research, Garden Grove, California
  - Synergy Escondido, La Mesa, California
  - Triwest Research Associates, La Mesa, California
  - LBCCR, Long Beach, California
  - Pacific Institute for Med Research, Los Angeles, California
  - Samaritan Center for Medical Research, Los Gatos, California
  - Synergy Research Center, National City, California
  - Northern California Research, Sacramento, California
  - Mountain View Clinical Research, Denver, Colorado
  - Avail Clinical Research, DeLand, Florida
  - Neuropsychiatric Research Center of SW Florida, Fort Myers, Florida
  - CNS Healthcare, Jacksonville, Florida
  - Florida Institute of Medical Research, Jacksonville, Florida
  - Behavioral Clinical Research, Inc., Lauderhill, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - CNS Health, Orlando, Florida
  - Compass Research, Orlando, Florida
  - Altas Orthopedics & Sports Medicine, Orlando, Florida
  - Gold Coast Research LLC., Plantation, Florida
  - Medex Healthcare Research, Inc., Chicago, Illinois
  - Center for Pain Management Rehabilitation Institute of Chicago, Chicago, Illinois
  - Integrated Clinical Trial Services Inc., West Des Moines, Iowa
  - International Clinical Research Institute Inc., Overland Park, Kansas
  - Robert Wagner, MD, Crestview Hills, Kentucky
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Beacon Clinical Research LLC, Brockton, Massachusetts
  - Quest Research Institute, Bingham Farms, Michigan
  - Prime Care Research Associates, Florissant, Missouri
  - Medex Health Research, Inc., St Louis, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Office of Danka Micheals, MD, Las Vegas, Nevada
  - Stephen Miller, MD, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Finger Lakes Clinical Research, Rochester, New York
  - New Hanover Medical Research, Wilmington, North Carolina
  - The Center for Clinical Research, LLC & Carolinas Pain Institute, P.A., Winstom-Salem, North Carolina
  - David Schneider, MD, Cincinnari, Ohio
  - Community Research, Cincinnati, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - Bone, Joint & Spine Surgeons, Inc., Toledo, Ohio
  - Neurology & Neruoscience Center of Ohio, Toledo, Ohio
  - Alleghany Pain Management, PC, Altoona, Pennsylvania
  - Paragon Clinical Research Inc., Cranston, Rhode Island
  - Omega Clinical Research, Warwick, Rhode Island
  - Future Search Trials, Ausitn, Texas
  - Austin Diagnostic Clinic, Ausitn, Texas
  - KRK Medical Research, Dallas, Texas
  - Clinical Trial Network, Houston, Texas
  - Medex Healthcare Research, Houston, Texas
  - Sun Research Institute, San Antonio, Texas